CLINICAL TRIAL: NCT07229040
Title: A Double-blind Non Inferiority Clinical Trial to Compare the Nephroprotection of Cilastatn Versus Thiosulfate in Patients Undergoing Debulking Surgery With Intraoperative Hyperthermic Intraperitoneal Chemotherapy With Cisplatin.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FIBHGM-ECNC001-2022; 2024-518854-18-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Debulking Surgery for Ovarian Cancer; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Cilastatin

STUDY DESIGN:
Intervention Model Description: Non inferiority study of cilastatin versus Thiosulfate
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cilastatin (Experimental): cilastatina 1,5 g
  Interventions: Drug: cilastatine
- tiosulfate (Active Comparator): tiosulfate
  Interventions: Drug: tiosulfate

INTERVENTIONS:
Drug: cilastatine — cilastatine 1.5 g
  Arms: cilastatin
Drug: tiosulfate — tiosulfate
  Arms: tiosulfate

SUMMARY:
To compare cilastatin vs thiosulfatein renal protection in patients undergoing debulking surgery with intraoperative hyperthermic intraperitoneal chemotherapy with cisplatin

DETAILED DESCRIPTION:
A double-blind non inferiority clinical trial to compare the nephroprotection of cilastatn versus thiosulfate in patients undergoing debulking surgery with intraoperative hyperthermic intraperitoneal chemotherapy with cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Age: adult patients aged 18-75 years.

Sex: female. Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 2. General condition: patients eligible for major surgery, with creatinine, bilirubin, and blood count values within or close to the normal range (Hb >10 g/dL, leukocytes >3,000/mL, neutrophils >1,000/mL, platelets >100,000/mL).

Patients evaluated by the Anesthesiology Department and deemed fit for surgery. Signed informed consent. Disease confined to the abdomen: CRS + HIPEC is not indicated in patients with pulmonary, bone, or other distant metastases. Patients with limited hematogenous metastases to the spleen or liver may be considered. Patients with regional or distant intra-abdominal lymphatic dissemination may also be considered, provided complete resection is feasible. FIGO stage IVA epithelial ovarian carcinoma at presentation, due to pleural effusion with mediastinal lymph node or splenic metastases, is an indication for neoadjuvant chemotherapy; if response is achieved, CRS + HIPEC may subsequently be considered.

Multidisciplinary Committee evaluation: radiological PCI is assessed, and the likelihood of achieving complete cytoreduction is estimated to determine the indication for CRS + HIPEC.

Exclusion Criteria:

* Lack of consent to participate in the clinical trial. Eastern Cooperative Oncology Group Performance Status (ECOG PS) > 2. Not eligible for major surgery. Disease not confined to the abdomen, or with findings indicating that optimal cytoreduction is not achievable (e.g., intestinal obstruction, biliary obstruction, ureteral obstruction, or diffuse involvement of the small bowel or mesentery).

Known hypersensitivity to platinum-based agents.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2028-10-21 (Estimated); Study Completion 2028-10-21 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with renal failure at 7 days | 7 days
  Percentage of patients with renal failure at 7 days (If renal impairment is present, follow-up continues until postoperative day 14), assessed based on serum creatinine levels and KDIGO classification criteria.
  Renal failure is defined as an increase in serum creatinine to 1.5-1.9 times the baseline value, or an increase in serum creatinine by ≥0.3 mg/dL (≥26.5 µmol/L), or a reduction in urine output to <0.5 mL/kg/hour for 6 to 12 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Hodpsital General Universitario Gregorio Marañón, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided